CLINICAL TRIAL: NCT01851967
Title: Effectiveness and Acceptability of MoodGYM in Treating Depressive Symptoms in Chinese Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Albert Yeung, Principle Investigator / Psychiatrist, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-P-002340
Record Dates: First submitted 2013-01-08; First posted 2013-05-13 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Major Depressive Disorder
Keywords: Major depressive disorder; Cognitive behavioral therapy; Computerized CBT; Online CBT
MeSH Terms: conditions — Depressive Disorder, Major

ARMS (1):
- MoodGYM (Experimental): This study is a single-arm intervnetion. All subjects will be assigned to receive six weeks of online CBT through MoodGYM.
  Interventions: Other: MoodGYM

INTERVENTIONS:
Other: MoodGYM — MoodGYM, a publicly-available online CBT program developed by the Centre for Mental Health Research at The Australian National University has been shown by multiple studies to be effective in reducing symptoms of depression. MoodGYM consists of five interactive modules. Participants will be asked to complete one module each week and progress through the program sequentially.

SUMMARY:
This study aims to evaluate efficacy and acceptability of the Chinese language version of MoodGYM as a therapeutic intervention in treating symptoms of depression in community dwelling Chinese Americans in the Boston area.

Hypothesis 1: Participants enrolled in MoodGYM will show a significant decrease in depressive symptoms after completion of the 5 modules.

Hypothesis 2: Participants enrolled in MoodGYM will show significantly improved dysfunctional thinking.

Hypothesis 3: Participants enrolled in MoodGym will rate this program as culturally acceptable.

ELIGIBILITY:
Inclusion Criteria:

* Resident of the US, but self-identified as Chinese origin
* At least 18 years of age
* Proficiency in Chinese, including the ability to read Chinese
* Access to computer and internet
* Scores > 10 on the Chinese bilingual patient health questionnaire -9 item (PHQ-9)

Exclusion Criteria:

* Current ongoing psychiatric or psychological treatment
* Using illicit drugs or consumption > 3 standard drinks in a day
* Currently experiencing a psychotic illness
* Past or current history of schizophrenia or bipolar disorder
* ECT during the last year
* Current active suicidal or self-injurious potential necessitating immediate face-to-face treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change in Center for Epidemiologic Studies Depression Scale (CES-D) | Weeks 0, 6 (pre/post)
  The CES-D scale is a short self-report scale designed to measure depressive symptomatology in the general population. Each of the 20 items in this instrument is assigned one value of 0, 1, 2 or 3. High scores on the CES-D indicate high levels of distress.

CONTACTS AND LOCATIONS:
Locations (2):
- Massachusetts General Hospital Depression Clinical and Research Program, Boston, Massachusetts, United States
- Ying Wang, Beijing, China